CLINICAL TRIAL: NCT02494986
Title: An Open-label, Roll-over Study With Rilpivirine in Combination With a Background Regimen Containing Other Antiretrovirals (ARVs) in Human Immunodeficiency Virus Type 1 (HIV-1) Infected Subjects Who Participated in Rilpivirine Pediatric Studies
Brief Title: A Roll-over Study With Rilpivirine for Human Immunodeficiency Virus Type 1 (HIV-1) Infected Participants Who Participated in Rilpivirine Pediatric Studies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107451; TMC278IFD3004 (Other: Janssen Research & Development, LLC); 2014-002471-28 (EudraCT Number); 2024-512889-33-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Human immunodeficiency virus type 1; Rilpivirine; Roll-over study; Pediatrics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Rilpivirine (Experimental): Participants will continue to receive oral tablets of rilpivirine (RPV) 25 milligram once daily (mg qd) or a weight-adjusted dose, in combination with an investigator selected background regimen consisting of other antiretrovirals (ARVs).
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Rilpivirine — Participants will continue to receive oral tablets of rilpivirine (RPV) 25 milligram once daily (mg qd) or a weight-adjusted dose, in combination with an investigator selected background regimen consisting of other ARVs.
  Other Names: TMC278, R278474

SUMMARY:
The purpose of this study is to provide continued access to rilpivirine (RPV) for participants who were treated with RPV in a clinical development pediatric study with rilpivirine and who, at the time of roll-over, experience and are expected to continue experiencing clinical benefit from RPV treatment.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (more than one hospital or clinical site work on a study), roll-over study to provide continued access to RPV for human immunodeficiency virus type 1 (HIV-1) infected participants. All enrolled participants will continue to receive RPV in combination with an investigator-selected background regimen consisting of other antiretrovirals (ARVs). Participants will continue to receive RPV in this study until one of the following criteria is met (whichever comes first) as determined in the study protocol: they meet at least one of the withdrawal criteria, or the participant has been treated in this roll-over study for 4 years (48 months) or older than 12 years of age and can continue RPV treatment outside of this roll-over study by switching to locally available RPV (if commercially available and reimbursed, or accessible through another source [example: access program or government program]) or other locally available RPV-based regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participants (or their legally acceptable representative) must sign an Informed Consent Form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. Assent is also required of children capable of understanding the nature of the study (typically 7 years of age and older)
* Participants must be human immunodeficiency virus type 1 (HIV-1) infected and must have previously been treated with rilpivirine (RPV) 25 mg qd (or weight-adjusted dose) in a clinical development pediatric study and completed the protocol-defined treatment period
* Participants must benefit from treatment with RPV, according to the efficacy and safety criteria as set out in the protocol of the pediatric study with RPV the participant was participating in prior to this rollover study, and must be expected to continue to benefit from this treatment in the opinion of the investigator
* Participants must be able and willing to comply with the current protocol requirements
* Participants' general medical condition, in the opinion of the investigator, does not interfere with participation in this study

Exclusion Criteria:

* Participants using disallowed concomitant treatment
* Pregnant participants
* Female participants of childbearing potential and non-vasectomized heterosexually active male participants not willing to continue practicing birth control methods during the study and for greater than or equal to (≥)1 month after the end of the study (or after last intake of RPV)
* Participants who were withdrawn from a pediatric study with RPV that they were participating in prior to this rollover study, based on any of the mandatory withdrawal criteria

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) related to rilpivirine (RPV) | Up to 32 Days from the last dose administered (Approximately 16 years)
  Evaluation of long term safety of the treatment with RPV with a background regimen. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with AEs Leading to Discontinuation | Up to 32 Days from the last dose administered (Approximately 16 years)
  Number of participants with AEs leading to discontinuation will be reported. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Serious Adverse Events (SAEs) | Up to 32 Days from the last dose administered (Approximately 16 years)
  Number of participants with SAEs will be reported. An SAE is any adverse event (AE) that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants with Pregnancies | Up to 32 Days from the last dose of administered (Approximately 16 years)
  Number of participants with pregnancies will be reported.
Number or Participants with Grade 3/4 Rash Regardless of Causality | Up to 32 Days from the last dose administered (Approximately 16 years)
  Number of participants with grade 3/4 rash regardless of causality will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trials, Study Director — Janssen R&D Ireland
Locations (8):
- Porto, Portugal
- South Africa (2):
  - Bloemfontein
  - Dundee
- Esplugues de Llobregat, Spain
- Thailand (2):
  - Bangkok
  - Nonthaburi
- Uganda (2):
  - Entebbe
  - Kampala